CLINICAL TRIAL: NCT01760317
Title: Midline vs Lateral Parasagittal Approach During Fluoroscopically Guided Interlaminar Lumbar Epidural Steroid Injection: the Role of Concordant Pressure Paresthesia in Determing Outcome.
Brief Title: Two Different Approaches During Fluoroscopically Guided Interlaminar Lumbar Epidural Steroid Injection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kenneth D Candido (Other)
Responsible Party: Sponsor-Investigator, Kenneth D Candido, Chairman of Anesthesia Department; Advocate Illinois Masonic Medical Center, Chicago Anesthesia Pain Specialists
Organization: Chicago Anesthesia Pain Specialists (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Advocate-IRB-4917
Record Dates: First submitted 2012-12-21; First posted 2013-01-04 (Estimated); Last update posted 2015-02-05 (Estimated); Status verified 2015-02

CONDITIONS: Unilateral Lumbosacral Radiculopathy Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Midline (Active Comparator): Midline Lumbar Epidural Steroid Injection
  Interventions: Procedure: Midline vs Parasagittal Lumbar Epidural Steroid Injection
- Parasagittal (Active Comparator): Parasagittal Lumbar Epidural Steroid Injection
  Interventions: Procedure: Midline vs Parasagittal Lumbar Epidural Steroid Injection

INTERVENTIONS:
Procedure: Midline vs Parasagittal Lumbar Epidural Steroid Injection

SUMMARY:
The purpose of this study is to compare two different approaches (midline and parasagittal) during interlaminar lumbar epidural steroid injection (LESI), and to verify the role of concordant pressure paresthesia occurring during the LESI in determining outcome.

The investigators are planning to include 100 patients, undergoing LESI for radicular low back pain. This will be single-blinded randomized study. Every patient will receive the same medication we would use regardless of participating in the study. The patients will be randomly assigned to one of two groups, based on the approach:

* Group I (50 patients) - will get LESI using midline (MIL) approach.
* Group II (50 patients) - will get LESI using parasagittal interlaminar (PIL) approach.

ELIGIBILITY:
Inclusion Criteria:

* 18- 80 years old
* History of low back pain and unilateral lumbosacral radiculopathy pain
* Lumbar disk disease including disk herniations, bulging discs, and degenerated discs, where at least 50% of the disk height is preserved respective to contiguous levels

Exclusion Criteria:

* Discogenic pain without radiculopathy pain
* History of previous spinal surgery
* LESI(s) in the past year
* Allergy to methylprednisolone, or lidocaine, or iodine-based contrast
* Concurrent use of systemic steroid medications
* Opioid habituation
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2010-08; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Changes in Pain Scores from baseline after Lumbar Epidural Steroid Injection | Days 1, 7, 14, 21, 28, 60, 120, 180, 360
Pressure Paresthesia during injection | 1 day (During Lumbar Epidural Steroid Injection)
Quality of life improvement change after Lumbar Epidural Steroid Injection | Days 1, 7, 14, 21, 28, 60, 120, 180, 360

CONTACTS AND LOCATIONS:
Locations (1):
- Chicago Anesthesia Pain Specialits, Chicago, Illinois, United States

REFERENCES:
- [Background] Boswell MV, Shah RV, Everett CR, Sehgal N, McKenzie Brown AM, Abdi S, Bowman RC 2nd, Deer TR, Datta S, Colson JD, Spillane WF, Smith HS, Lucas LF, Burton AW, Chopra P, Staats PS, Wasserman RA, Manchikanti L. Interventional techniques in the management of chronic spinal pain: evidence-based practice guidelines. Pain Physician. 2005 Jan;8(1):1-47. PMID 16850041
- [Background] Abdi S, Datta S, Trescot AM, Schultz DM, Adlaka R, Atluri SL, Smith HS, Manchikanti L. Epidural steroids in the management of chronic spinal pain: a systematic review. Pain Physician. 2007 Jan;10(1):185-212. PMID 17256030
- [Background] Manchikanti L. The growth of interventional pain management in the new millennium: a critical analysis of utilization in the medicare population. Pain Physician. 2004 Oct;7(4):465-82. PMID 16858489
- [Background] Boswell MV, Trescot AM, Datta S, Schultz DM, Hansen HC, Abdi S, Sehgal N, Shah RV, Singh V, Benyamin RM, Patel VB, Buenaventura RM, Colson JD, Cordner HJ, Epter RS, Jasper JF, Dunbar EE, Atluri SL, Bowman RC, Deer TR, Swicegood JR, Staats PS, Smith HS, Burton AW, Kloth DS, Giordano J, Manchikanti L; American Society of Interventional Pain Physicians. Interventional techniques: evidence-based practice guidelines in the management of chronic spinal pain. Pain Physician. 2007 Jan;10(1):7-111. PMID 17256025
- [Background] Buenaventura RM, Datta S, Abdi S, Smith HS. Systematic review of therapeutic lumbar transforaminal epidural steroid injections. Pain Physician. 2009 Jan-Feb;12(1):233-51. PMID 19165306
- [Background] Candido KD, Raghavendra MS, Chinthagada M, Badiee S, Trepashko DW. A prospective evaluation of iodinated contrast flow patterns with fluoroscopically guided lumbar epidural steroid injections: the lateral parasagittal interlaminar epidural approach versus the transforaminal epidural approach. Anesth Analg. 2008 Feb;106(2):638-44, table of contents. doi: 10.1213/ane.0b013e3181605e9b. PMID 18227326